CLINICAL TRIAL: NCT01120093
Title: Efficacy and Safety of Three Doses of Aclidinium Bromide Compared to Placebo and to an Active Comparator All Administered Twice Daily by Inhalation in Patients With Stable Moderate and Severe Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Efficacy and Safety of Three Doses of Aclidinium Bromide Compared to Placebo and to an Active Comparator in Chronic Obstructive Pulmonary Disease (COPD) Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M/34273/29; LAS29
Record Dates: First submitted 2010-05-07; First posted 2010-05-10 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; BID protein, human; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Aclidinium bromide 100 μg bid (Experimental): Aclidininum bromide 100 μg twice daily by inhalation
  Interventions: Drug: Aclidinium bromide 100 μg bid
- Aclidininum bromide 200 μg bid (Experimental): Aclidininum bromide 200 μg twice daily by inhalation
  Interventions: Drug: Aclidinium bromide 200 μg bid
- Aclidininum bromide 400 μg bid (Experimental): Aclidininum bromide 400 μg twice daily by inhalation
  Interventions: Drug: Aclidininum bromide 400 μg bid
- Placebo (Placebo Comparator): Placebo twice-daily by inhalation
  Interventions: Drug: Placebo
- Formoterol 12 μg bid (Active Comparator): Formoterol 12 μg twice daily by inhalation
  Interventions: Drug: Formoterol 12 μg bid

INTERVENTIONS:
Drug: Aclidinium bromide 100 μg bid — Aclidinium bromide 100 μg twice-daily via inhalation by Eklira Genuair® inhaler: 1 puff in the morning and evening for 7 days
  Arms: Aclidinium bromide 100 μg bid
Drug: Aclidinium bromide 200 μg bid — Aclidinium bromide 200 μg twice-daily via inhalation by Eklira Genuair® inhaler: 1 puff in the morning and evening for 7 days
  Arms: Aclidininum bromide 200 μg bid
Drug: Aclidininum bromide 400 μg bid — Aclidinium bromide 400 μg twice-daily via inhalation by Eklira Genuair® inhaler: 1 puff in the morning and evening for 7 days
  Arms: Aclidininum bromide 400 μg bid
Drug: Placebo — Placebo via inhalation in the morning and evening for 7 days
  Arms: Placebo
Drug: Formoterol 12 μg bid — Formoterol 12 μg twice-daily via inhalation by Aerolizer® dry powder inhaler: 1 puff in the morning and evening for 7 days
  Arms: Formoterol 12 μg bid

SUMMARY:
The present trial is conducted to further assess the efficacy by means of serial spirometry, safety and tolerability of three doses of aclidinium bromide administered twice a day compared to previously approved BID drug, formoterol 12 µg, and placebo in patients with moderate to severe chronic obstructive pulmonary disease (COPD).after 7 days on treatment. Every treatment period is 7-days long and there is a 5 to 7-days wash-out period in between them. The trial starts with a run in phase of 11 to 17-days duration and it ends up with a follow up contact 14-days after last treatment dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females aged ≥ 40.
2. Patients with a clinical diagnosis of stable moderate to severe COPD, according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines: (http://www.goldcopd.com) and stable airway obstruction. Post-salbutamol FEV1/FVC < 70% at Screening Visit (Visit 1) (i.e., 100xpost-salbutamol FEV1/FVC <70%).
3. Current, or ex-cigarette smoker with a smoking history of at least 10 pack-years.
4. Patient whose FEV1 at the Screening Visit measured between 10-15 minutes post inhalation of salbutamol is 30% < FEV1 <80% of the predicted normal value (i.e., 100 x Post-salbutamol FEV1/ Predicted FEV1 must be < 80% and ≥ 30%).
5. Female patients at least 1 year post-menopausal, surgically sterile (defined as having a hysterectomy or tubal ligation), or practicing a medically approved and highly effective method of contraception.
6. Patients who understand the study procedures and are willing to participate in the study as indicated by signing the informed consent.

Exclusion Criteria:

1. History or current diagnosis of asthma.
2. Clinically significant respiratory conditions other than COPD at the time of Inform Consent signature
3. Hospitalisation due to COPD exacerbation within the previous 3 months.
4. Signs of a COPD exacerbation or respiratory infection (including the upper respiratory tract) within the previous 6 weeks.
5. Clinically significant cardiovascular conditions
6. Presence of symptomatic prostatic hypertrophy and/or bladder neck obstruction.
7. Presence of narrow-angle glaucoma.
8. QTcB) above 470 milliseconds in the ECG performed at Screening Visit,
9. Patient who does not maintain regular day/night, waking/sleeping cycles

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (11):
- Almirall Investigational Sites#1, Ghent, Belgium
- Germany (10):
  - Almirall Investigational Sites#3, Berlin
  - Almirall Investigational Sites#4, Berlin
  - Almirall Investigational Sites#9, Berlin
  - Almirall Investigational Sites#8, Frankfurt
  - Almirall Investigational Sites#1, Groβhansdorf
  - Almirall Investigational Sites#5, Hamburg
  - Almirall Investigational Sites#7, Hanover
  - Almirall Investigational Sites#2, Hanover
  - Almirall Investigational Sites#6, Schwerin
  - Almirall Investigational Sites#10, Wiesbaden

REFERENCES:
- [Derived] Singh D, Magnussen H, Kirsten A, Mindt S, Caracta C, Seoane B, Jarreta D, Garcia Gil E. A randomised, placebo- and active-controlled dose-finding study of aclidinium bromide administered twice a day in COPD patients. Pulm Pharmacol Ther. 2012 Jun;25(3):248-53. doi: 10.1016/j.pupt.2012.03.008. Epub 2012 Apr 4. PMID 22497752
- See also: Almirall Corporate Website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3977&filename=Synopsis_m-34273-29-Final.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a total of 11 centres; 10 in Germany and 1 in Belgium. The first patient was screened in Apr 2010 and the last patient visit was in Aug 2010.
Pre-assignment Details: Patients fulfilling inclusion/exclusion criteria at the time of the Screening Visit were entered into a run-in period of 14 ± 3 days to assess patient's disease stability.
Groups:
- Aclidinium100;Aclidinium200;Placebo;Aclidinium400;Formoterol: The treatment period consisted of 5 periods of 7 treatment days each separated by a washout period of 7 (±2) days.
  In period 1, patients received aclidinium bromide 100 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 2, patients received aclidinium bromide 200 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 3, patients received placebo from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 4, patients received aclidinium bromide 400 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 5, patients received placebo from the Eklira Genuair® inhaler and formoterol from the Aerolizer® inhaler in the morning and evening for 7 days.
- Aclidinium200;Aclidinium400;Aclidinium100;Formoterol;Placebo: The treatment period consisted of 5 periods of 7 treatment days each separated by a washout period of 7 (±2) days.
  In period 1, patients received aclidinium bromide 200 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 2, patients received aclidinium bromide 400 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 3, patients received aclidinium bromide 100 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 4, patients received placebo from the Eklira Genuair® inhaler and formoterol from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 5, patients received placebo from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
- Aclidinium400;Formoterol;Aclidinium200;Placebo;Aclidinium100: The treatment period consisted of 5 periods of 7 treatment days each separated by a washout period of 7 (±2) days.
  In period 1, patients received aclidinium bromide 400 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 2, patients received placebo from the Eklira Genuair® inhaler and formoterol from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 3, patients received aclidinium bromide 200 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 4, patients received placebo from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 5, patients received aclidinium bromide 100 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
- Formoterol;Placebo;Aclidinium400;Aclidinium100;Aclidinium200: The treatment period consisted of 5 periods of 7 treatment days each separated by a washout period of 7 (±2) days.
  In period 1, patients received placebo from the Eklira Genuair® inhaler and formoterol from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 2, patients received placebo from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 3, patients received aclidinium bromide 400 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 4, patients received aclidinium bromide 100 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 5, patients received aclidinium bromide 200 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
- Placebo;Aclidinium100;Formoterol;Aclidinium200;Aclidinium400: The treatment period consisted of 5 periods of 7 treatment days each separated by a washout period of 7 (±2) days.
  In period 1, patients received placebo from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 2, patients received aclidinium bromide 100 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 3, patients received placebo from the Eklira Genuair® inhaler and formoterol from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 4, patients received aclidinium bromide 200 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
  In period 5, patients received aclidinium bromide 400 μg from the Eklira Genuair® inhaler and placebo from the Aerolizer® inhaler in the morning and evening for 7 days.
Period: Treatment Period 1
Arm/Group | Aclidinium100;Aclidinium200;Placebo;Aclidinium400;Formoterol | Aclidinium200;Aclidinium400;Aclidinium100;Formoterol;Placebo | Aclidinium400;Formoterol;Aclidinium200;Placebo;Aclidinium100 | Formoterol;Placebo;Aclidinium400;Aclidinium100;Aclidinium200 | Placebo;Aclidinium100;Formoterol;Aclidinium200;Aclidinium400
Started | 18 | 14 | 17 | 14 | 16
Completed | 18 | 13 | 16 | 14 | 15
Not Completed | 0 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Aclidinium100;Aclidinium200;Placebo;Aclidinium400;Formoterol | Aclidinium200;Aclidinium400;Aclidinium100;Formoterol;Placebo | Aclidinium400;Formoterol;Aclidinium200;Placebo;Aclidinium100 | Formoterol;Placebo;Aclidinium400;Aclidinium100;Aclidinium200 | Placebo;Aclidinium100;Formoterol;Aclidinium200;Aclidinium400
Started | 18 | 13 | 16 | 14 | 15
Completed | 18 | 13 | 16 | 13 | 14
Not Completed | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 3
Arm/Group | Aclidinium100;Aclidinium200;Placebo;Aclidinium400;Formoterol | Aclidinium200;Aclidinium400;Aclidinium100;Formoterol;Placebo | Aclidinium400;Formoterol;Aclidinium200;Placebo;Aclidinium100 | Formoterol;Placebo;Aclidinium400;Aclidinium100;Aclidinium200 | Placebo;Aclidinium100;Formoterol;Aclidinium200;Aclidinium400
Started | 18 | 13 | 16 | 13 | 14
Completed | 18 | 13 | 15 | 12 | 13
Not Completed | 0 | 0 | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: Treatment Period 4
Arm/Group | Aclidinium100;Aclidinium200;Placebo;Aclidinium400;Formoterol | Aclidinium200;Aclidinium400;Aclidinium100;Formoterol;Placebo | Aclidinium400;Formoterol;Aclidinium200;Placebo;Aclidinium100 | Formoterol;Placebo;Aclidinium400;Aclidinium100;Aclidinium200 | Placebo;Aclidinium100;Formoterol;Aclidinium200;Aclidinium400
Started | 18 | 13 | 15 | 12 | 13
Completed | 17 | 13 | 15 | 12 | 13
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 5
Arm/Group | Aclidinium100;Aclidinium200;Placebo;Aclidinium400;Formoterol | Aclidinium200;Aclidinium400;Aclidinium100;Formoterol;Placebo | Aclidinium400;Formoterol;Aclidinium200;Placebo;Aclidinium100 | Formoterol;Placebo;Aclidinium400;Aclidinium100;Aclidinium200 | Placebo;Aclidinium100;Formoterol;Aclidinium200;Aclidinium400
Started | 17 | 13 | 15 | 12 | 13
Completed | 17 | 12 | 15 | 11 | 13
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All patients randomized into the crossover study
Arm/Group | Overall Study Population
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (8.5)
Gender [Count of Participants; unit: Participants]
  Female | 20
  Male | 59
Region of Enrollment [Number; unit: participants]
  Belgium | 3
  Germany | 76

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in First Second (FEV1) Area Under Curve (AUC) 0-12h at Day 7 on Treatment
Time Frame: Day 7
Population: Intention-to-treat (ITT) population; patients were included who took at least one dose of Investigational Medicinal Product and had at least a baseline and one post-dose value of FEV1
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Aclidinium Bromide 100 μg Bid: Aclidinium bromide 100 μg twice-daily via inhalation
- Aclidinium Bromide 200 μg Bid: Aclidinium bromide 200 μg twice-daily via inhalation
- Aclidinium Bromide 400 μg Bid: Aclidinium bromide 400 μg twice-daily via inhalation
- Formoterol 12 μg Bid: Formoterol 12 μg twice-daily via inhalation
- Placebo: Placebo via inhalation
Arm/Group | Aclidinium Bromide 100 μg Bid | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Formoterol 12 μg Bid | Placebo
Number analyzed (Participants) | 73 | 71 | 73 | 74 | 73
Liters | 0.128 (0.022) | 0.151 (0.022) | 0.183 (0.022) | 0.184 (0.022) | -0.026 (0.022)

2. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in First Second (FEV1) Area Under Curve (AUC) 12-24h at Day 7 on Treatment
Time Frame: Day 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 100 μg Bid | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Formoterol 12 μg Bid | Placebo
Number analyzed (Participants) | 72 | 69 | 71 | 72 | 72
Liters | 0.044 (0.021) | 0.047 (0.021) | 0.086 (0.021) | 0.141 (0.021) | -0.103 (0.021)

3. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in First Second (FEV1) Area Under Curve (AUC) 0-24h at Day 7 on Treatment
Time Frame: Day 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 100 μg Bid | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Formoterol 12 μg Bid | Placebo
Number analyzed (Participants) | 72 | 69 | 71 | 74 | 72
Liters | 0.088 (0.021) | 0.100 (0.021) | 0.133 (0.021) | 0.163 (0.021) | -0.062 (0.021)

4. Secondary Outcome: Change From Baseline in Morning Pre-dose Forced Expiratory Volume in First Second (FEV1) at Day 7 on Treatment
Time Frame: Day 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 100 μg Bid | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Formoterol 12 μg Bid | Placebo
Number analyzed (Participants) | 73 | 72 | 73 | 74 | 75
Liters | 0.081 (0.023) | 0.089 (0.023) | 0.130 (0.023) | 0.123 (0.023) | -0.025 (0.023)

ADVERSE EVENTS:
Groups:
- Aclidinium Bromide 100 μg Bid: Aclidinium bromide 100 μg twice-daily via inhalation by Genuair® multidose dry powder inhaler: 1 puff at 09:00 (± 30 mins) and at 21:00 (± 30 mins) for 7 days.
- Aclidinium Bromide 200 μg Bid: Aclidinium bromide 200 μg twice-daily via inhalation by Genuair® multidose dry powder inhaler: 1 puff at 09:00 (± 30 mins) and at 21:00 (± 30 mins) for 7 days.
- Aclidinium Bromide 400 μg Bid: Aclidinium bromide 400 μg twice-daily via inhalation by Genuair® multidose dry powder inhaler: 1 puff at 09:00 (± 30 mins) and at 21:00 (± 30 mins) for 7 days.
- Formoterol 12 μg Bid: Formoterol 12 μg twice-daily via inhalation by Aerolizer® inhaler at 09:00 (± 30 mins) and 21:00 (± 30 mins) for 7 days.
- Placebo: Inhaled placebo dose for 7 days.
Arm/Group | Aclidinium Bromide 100 μg Bid | Aclidinium Bromide 200 μg Bid | Aclidinium Bromide 400 μg Bid | Formoterol 12 μg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/73 | 1/73 | 1/74 | 0/74 | 2/76
Other Adverse Events (participants affected / at risk) | 4/73 | 4/73 | 5/74 | 2/74 | 1/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide 100 μg Bid (N=73) | Aclidinium Bromide 200 μg Bid (N=73) | Aclidinium Bromide 400 μg Bid (N=74) | Formoterol 12 μg Bid (N=74) | Placebo (N=76)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious exacerbation of chronic obstructive pulmonary disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium Bromide 100 μg Bid (N=73) | Aclidinium Bromide 200 μg Bid (N=73) | Aclidinium Bromide 400 μg Bid (N=74) | Formoterol 12 μg Bid (N=74) | Placebo (N=76)
Headache (Nervous system disorders) | 4 | 4 | 5 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of Almirall. This information will not be given to a third party without the written consent of Almirall. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and Almirall.